CLINICAL TRIAL: NCT03411447
Title: Impact of Early Enteral vs. Parenteral Nutrition on Risk of Gastric-Content Aspiration in Patients Requiring Mechanical Ventilation and Catecholamines: an Ancillary Study of the NUTRIREA2 Trial (NCT01802099)
Brief Title: Impact of Early Enteral vs. Parenteral Nutrition on Risk of Gastric-Content Aspiration in Patients Requiring Mechanical Ventilation and Catecholamines
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped on Data Safety and Monitoring Board 's request
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD085-13
Record Dates: First submitted 2017-07-18; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Acute Respiratory Failure; Shock
Keywords: vasoactive drug; mechanical ventilation; early enteral nutrition; intensive care unit; early parenteral nutrition; critical care medicine; nosocomial infection; mortality; shock
MeSH Terms: conditions — Shock; Hyperphagia; Cross Infection | interventions — Parenteral Nutrition; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenteral nutrition (Active Comparator): Patients will receive parenteral nutrition during the first week of mechanical ventilation. After Day 3, the parenteral route may be switched to the enteral route if shock resolve (vasoactive drug stopped since 24 hours and serum lactate level < 2 mmol/l). After Day 7, all patients will be fed via the enteral route.
  Interventions: Other: Parenteral nutrition
- Enteral nutrition (Active Comparator): Patients will receive nutrition only via the enteral route during the firs week of invasive mechanical ventilation.
  Interventions: Other: Enteral nutrition

INTERVENTIONS:
Other: Parenteral nutrition
  Other Names: Intravenous nutrition; Intravenous feeding
  Arms: Parenteral nutrition
Other: Enteral nutrition
  Other Names: Enteral feeding
  Arms: Enteral nutrition

SUMMARY:
To evaluate the impact of enteral nutrition on microaspiration of gastric content and pharyngeal secretions

DETAILED DESCRIPTION:
A common obstacle to enteral nutrition is gastrointestinal intolerance, with regurgitations potentially responsible for gastric-content aspiration. Several studies involving technetium 99m (99mTc) labeling of gastric contents have established that gastric-fluid microaspiration is common in critically ill patients receiving both endotracheal ventilation and enteral nutrition. However, to our knowledge, no studies have specifically addressed the role for enteral nutrition in the occurrence of microaspiration. The objective of this ancillary study is to compare the frequency of gastric-content microaspiration in patients given enteral versus parenteral nutrition during the NUTRIREA2 trial. The new knowledge of risk factors for microaspiration provided by this study may help to improve strategies for preventing microaspiration and ventilator-associated pneumonia (VAP).

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation expected to be required more than 48 hours
* Nutrition started within 24 hours after initiation of endotracheal mechanical ventilation
* Treatment with vasoactive drug administered via a central venous catheter
* Age over 18 years
* Signed information

Exclusion Criteria:

* Abdominal surgery within 1 month before inclusion
* History of esophageal, gastric, duodenal or pancreatic surgery
* Bleeding from the esophagus, stomach or bowel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
proportion of patients with abundant microaspiration (defined as a pepsin level >200 ng/mL in at least 30% of tracheal aspirates) | 48Hours following randomisation
  Every tracheal aspirate will be collected during 48hours following randomisation

SECONDARY OUTCOMES:
Salivary amylase levels in tracheal aspirates. | 48Hours following randomisation
  Every tracheal aspirate will be collected during 48hours following randomisation. Salivary amylase will be analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Jean REIGNIER, MD, PhD, Principal Investigator — CHD Vendee
Locations (6):
- France (6):
  - CHU Amiens, Amiens
  - Centre hospitalier d'Annecy, Annecy
  - CHU Louis Mourier, Colombes
  - CHU Lille, Lille
  - CHU Saint Louis, Paris
  - CHU Tours, Tours

REFERENCES:
- [Derived] Nseir S, Le Gouge A, Lascarrou JB, Lacherade JC, Jaillette E, Mira JP, Mercier E, Declercq PL, Sirodot M, Piton G, Tinturier F, Coupez E, Gaudry S, Djibre M, Thevenin D, Pasco J, Balduyck M, Zerimech F, Reignier J. Impact of nutrition route on microaspiration in critically ill patients with shock: a planned ancillary study of the NUTRIREA-2 trial. Crit Care. 2019 Apr 5;23(1):111. doi: 10.1186/s13054-019-2403-z. PMID 30953553